CLINICAL TRIAL: NCT01402206
Title: Management of Depression in Primary Health Care: a Controlled Trial on the Effectiveness of Regular, Structured, Patient-centered Visits
Brief Title: Management of Depression in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Madrs 2010
Record Dates: First submitted 2011-06-27; First posted 2011-07-26 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: Depression; Intervention; Primary health care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured patient visits (Other): Participants in the intervention group visit their general practitioner at baseline and 4, 8, and 12 weeks. At each visit, participants complete MADRS-s for the assessment of depression severity and discuss the results with their GP in a patient-centered consultation.
  Interventions: Behavioral: Structured patient-centered follow up of depression
- Treatment as usual (Other): The control group receives treatment as usual by general practitioner (no intervention).
  Interventions: Behavioral: Structured patient-centered follow up of depression

INTERVENTIONS:
Behavioral: Structured patient-centered follow up of depression — All patients who agree to participate in the study are diagnosed by their GP with a diagnostic assessment instrument called PRIME-MD. Participants in the intervention group visit their GPs at baseline and 4, 8, and 12 weeks. At each visit, participants complete MADRS-s for the assessment of depression severity and discuss the results with their GP in a patient-centered consultation. We have chosen to use the MADRS/MADRS-S depression rating scale in this study because it is a easy to use standard instrument especially suitable for measuring change in depressive symptoms.
  The control group receives treatment as usual (no intervention).
  Other Names: MADRS/MADRS-S depression rating scale

SUMMARY:
Most people in Sweden with mild to moderate depression are treated in primary care, but follow-up is unstructured, and we know little about whether structured, follow-up would affect the prognosis for depression and working life. The purpose of this study is to determine the effectiveness of regular, structured, patient-centered visits on mild to moderate depression.

ELIGIBILITY:
Inclusion criteria

* Age 18 years and up
* Attends a participating primary health care center in the region
* Diagnosis of mild/moderate depressive disorder (new episode)
* No change in possible antidepressant maintenance therapy during the preceding 1 month
* Provided written informed consent

Exclusion criteria

* Antidepressant medication initiated or changed during the preceding 1 month
* Patient diagnosed with major depressive disorder (BDI-II >28)
* Patients diagnosed of severe mental psychiatric disorder (i.e. bipolar disorder, antisocial personality disorder, psychosis, substance use disorder or other serious mental disorder)
* Suicidal ideation or intentions
* Inability to speak and understand Swedish language well enough to take part in the activities required in the study.
* Cognitive impairment that makes it impossible to take part in the activities required in the study
* Does not provide written informed consent to participation in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Depressive symptoms | 3, 6 and 12 months.
  Depressive symptoms will be assessed using the Beck Depression Inventory (BDI-II), a self-administered questionnaire that measures the symptoms and severity of the depression.

SECONDARY OUTCOMES:
Change in Quality of life | 3, 6 and 12 months
  Each patient's quality of life will be assessed using the EuroQoL-5D questionnaire that measures five dimensions of quality of life
Prescriptions for antidepressants | 12-month follow-up period
  Information on Antidepressant use will be collected from patient records from start of the study and the 12-month follow-up period
Change in Activity/work ability | 12-month follow-up period
  Will be measured by Work Ability Index (WAI) and the Karaseks Job Strain Model Questionnaire. The Work Ability Index is used for evaluating people's work capacity and Karaseks Job Strain Model Questionnaire is used for evaluating Demands-Control in work place
sick-listing data | 12 month follow up
  Data on sick-listing is derived from primary care record fom baseline to 3 months follow up and from patient interview from 3 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cecila Björkelund, Professor, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Wikberg C, Westman J, Petersson EL, Larsson ME, Andre M, Eggertsen R, Thorn J, Agren H, Bjorkelund C. Use of a self-rating scale to monitor depression severity in recurrent GP consultations in primary care - does it really make a difference? A randomised controlled study. BMC Fam Pract. 2017 Jan 19;18(1):6. doi: 10.1186/s12875-016-0578-9. PMID 28103816